CLINICAL TRIAL: NCT03112772
Title: Socket Preservation for Dental Implant Site Development.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imam Abdulrahman Al Faisal Hospital (Other Government)
Responsible Party: Principal Investigator, Hesham Marei, Associate professor and Consultant of Oral and Maxillofacial Surgery, Imam Abdulrahman Al Faisal Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014342
Record Dates: First submitted 2017-04-08; First posted 2017-04-13 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (Experimental): Participants who are receiving socket preservation using allograft (Puros® Allograft, Zimmer dental, Zimmer, USA) covered by membrane (size: 15x20mm) made of type I collagen fibers purified from bovine tendon (BioMend® Membrane, Zimmer dental, Zimmer, USA).
  Interventions: Other: Puros® Allograft
- Group II (Experimental): Participants who are receiving socket preservation cancellous particulate bovine bone xenograft (CopiOs® Cancellous Particulate, Zimmer dental, Zimmer, USA) covered by membrane (size: 15x20mm) made of type I collagen fibers purified from bovine tendon (BioMend® Membrane, 15x20mm, Zimmer dental, Zimmer, USA).
  Interventions: Other: CopiOs® Cancellous Particulate
- Group III (No Intervention): No grafting materials will be inserted, so it serves as a negative control group.

INTERVENTIONS:
Other: Puros® Allograft — It is a type of bone grafting materials used for enhancing bone formation
  Arms: Group I
Other: CopiOs® Cancellous Particulate — It is a type of bone grafting materials used for enhancing bone formation
  Arms: Group II

SUMMARY:
Changes in alveolar bone following teeth extraction can compromise implant placement. Socket preservation (alveolar ridge preservation) is considered as a surgical procedure employed to preserve the ridge volume within the envelope existing at the time of extraction.The ultimate aim of such procedure is to compensate the expected amount of horizontal and vertical alveolar bone resorption. In order to better understand which socket preservation materials might be more effective for ridge preservation and to strengthen the evidence that is relevant to the clinicians' choice of socket preservation materials, two different materials were compared in a randomized controlled approach. (1) Demineralized Bone Matrix (DBM) Putty and Putty with Chips allograft covered by collagen membrane, and (2) Deprotonated bovine bone xenograft covered by collagen membrane. The independent variable is the grafting material while the dependent variables are the change in socket height, and width; the ability of implant placement without the need for grafting and the success rate of implants at the time of loading.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient > 18 years old.
2. Single and or multi-rooted teeth that are non-restorable.
3. Patients are keen to have implant placement at the extraction sites after 4 months of extraction.
4. Intact buccal bone after extraction, which was confirmed by visual inspection and clinical examination using a periodontal probe.
5. Patients are medically fit with no underlying systemic diseases.

Exclusion Criteria:

1. Pregnant females.
2. Smokers.
3. Presence of any acute infection at the time of teeth extraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-07-20 (Estimated); Study Completion 2017-11-20 (Estimated)

PRIMARY OUTCOMES:
Width of alveolar ridge | 4 months
  The distance from the buccal to the lingual surface of the alveolar ridge
height of the alveolar ridge | 4 months
  The distance from the crest of the ridge to the base of the socket
Need of further grafting at the time of implant placement | 4 months
  Ability to place implants

SECONDARY OUTCOMES:
Osseintegration of implants | 4 months
  Implant loss before restoration

CONTACTS AND LOCATIONS:
Locations (1):
- Immam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after statistical analysis